CLINICAL TRIAL: NCT04695392
Title: Restore Resilience in Critically Ill Children
Acronym: R2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Johns Hopkins University (Other); Children's Hospital of Philadelphia (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Martha A.Q. Curley, PhD, RN, Principal Investigator, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 828061
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): R2 Bundle
  Interventions: Other: R2 Bundle
- Baseline (No Intervention): Usual care

INTERVENTIONS:
Other: R2 Bundle — During the intervention phase subjects will receive R2.
  1. Focused effort to replicate the child's pre-hospitalization daily routine (bedtime/wake time, bedtime/arousal routine, nap time, feeding schedule, active periods),
  2. Cycled day-night lighting and modulation of sound to match the child's routine,
  3. Minimal yet effective sedation using a nurse-implemented goal-directed sedation plan (RESTORE),
  4. Night fasting with bolus enteral daytime feedings,
  5. Early, developmentally-appropriate, progressive exercise and mobility (PICU Up!),
  6. Continuity in nursing care, and
  7. Parent diaries.
  Arms: Intervention

SUMMARY:
The study design will allow investigators to describe usual care in each PICU and identify the facilitating and restraining factors impacting the implementation of R2 at each PICU. The purpose of this pilot study is to improve the care, environment, daily routine and sleep patterns of children in the PICU. The goal of this study is to learn what can be improved to support a critically ill child's healing and circadian rhythms.

DETAILED DESCRIPTION:
Hospitals should do the sick no harm. That noted, modern day pediatric intensive care units (PICUs) are not healing milieus. Immediately upon admission to the PICU, the child's daily routine and sleep patterns are replaced by a well-intended but not patient-centered PICU routine. The interprofessional investigative team believes that PICU care and environments can be modulated to sustain a young child's circadian rhythm (CR) and support their physiological resilience and capacity to heal. The first step in this program of research is to pilot-test RESTORE resilience (R2), a 7-item individualized bundle that we hypothesize will restore CR in critically ill children using a pre-posttest design. Two separate PICUs will each enroll 10 baseline subjects followed by 20 intervention subjects, 6 months to 18 years of age, who are intubated and mechanically ventilated for acute respiratory failure. Specifically, as soon as possible after PICU admission, parents will be interviewed to create an individualized chronotherapeutic bundle to include (1) focused effort to replicate the child's pre-hospitalization daily routine (bedtime/wake time, bedtime/arousal routine, nap time, feeding schedule, active periods), (2) cycled day-night lighting and modulation of sound to match the child's routine, (3) minimal yet effective sedation using a nurse-implemented goal-directed sedation plan (RESTORE), (4) night fasting with bolus enteral daytime feedings, (5) early, developmentally-appropriate, progressive exercise and mobility (PICU Up!), (6) continuity in nursing care, and (7) parent diaries. The overall objective of this study is to pilot-test an intervention that can be implemented in any PICU that will improve sleep-wake patterns with restoration/maintenance of circadian rhythms in critically ill children with acute respiratory failure. Results of this pilot study will be used to inform the design of an adequately powered multicenter randomized trial of R2.

ELIGIBILITY:
Inclusion Criteria:

* PICU admission at one of the study sites in which elements of R2 are typically but sporadically implemented
* Transferred to the PICU from another hospital unit/ward with ≤4 nights in the hospital (≤2 nights in PICU)
* Between the ages 6 months and 18 years at the time of enrollment (has not had their 18th birthday)
* Intubated and mechanically ventilated for acute airway or parenchymal disease within last 48 hours
* Expected to be intubated for more than 12 hours past enrollment
* Parent/Guardian providing consent, provides primary care for subject

Exclusion Criteria:

* A baseline cognitive dysfunction, measured by the Pediatric Cerebral Performance Category (PCPC ≥4)
* A history of an uncontrolled seizure disorder (seizure within past 3 months), cerebral hypertension, neuromuscular respiratory failure, ventilator dependence (excluding BiPAP or CPAP at night)
* A history of inability to tolerate bolus enteral feeds (full J-Tube fed patients)
* The presence of any of the following within 24 hours of admission:

  * Modal pain scores greater than 4
  * Persistent hypotension/hypertension unresponsive to standard therapies
  * Use of High Frequency Oscillatory Ventilation or Extracorporeal Membrane Oxygenation
* Administered melatonin within the past week
* Has an active do-not-resuscitate plan

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha AQ Curley, RN, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Johns Hopkins University - Charlotte Bloomberg Children's Center, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wieczorek B, Burke C, Al-Harbi A, Kudchadkar SR. Early mobilization in the pediatric intensive care unit: a systematic review. J Pediatr Intensive Care. 2015;2015(4):129-170. doi: 10.1055/s-0035-1563386. Epub 2015 Sep 3. PMID 26380147
- [Background] Pollack MM, Holubkov R, Funai T, Berger JT, Clark AE, Meert K, Berg RA, Carcillo J, Wessel DL, Moler F, Dalton H, Newth CJ, Shanley T, Harrison RE, Doctor A, Jenkins TL, Tamburro R, Dean JM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Simultaneous Prediction of New Morbidity, Mortality, and Survival Without New Morbidity From Pediatric Intensive Care: A New Paradigm for Outcomes Assessment. Crit Care Med. 2015 Aug;43(8):1699-709. doi: 10.1097/CCM.0000000000001081. PMID 25985385
- [Background] Pollack MM, Holubkov R, Funai T, Clark A, Berger JT, Meert K, Newth CJ, Shanley T, Moler F, Carcillo J, Berg RA, Dalton H, Wessel DL, Harrison RE, Doctor A, Dean JM, Jenkins TL; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Pediatric intensive care outcomes: development of new morbidities during pediatric critical care. Pediatr Crit Care Med. 2014 Nov;15(9):821-7. doi: 10.1097/PCC.0000000000000250. PMID 25226501
- [Background] Hopkins RO, Choong K, Zebuhr CA, Kudchadkar SR. Transforming PICU Culture to Facilitate Early Rehabilitation. J Pediatr Intensive Care. 2015 Dec;4(4):204-211. doi: 10.1055/s-0035-1563547. PMID 27134761
- [Background] Kamdar BB, Niessen T, Colantuoni E, King LM, Neufeld KJ, Bienvenu OJ, Rowden AM, Collop NA, Needham DM. Delirium transitions in the medical ICU: exploring the role of sleep quality and other factors. Crit Care Med. 2015 Jan;43(1):135-141. doi: 10.1097/CCM.0000000000000610. PMID 25230376
- [Background] Gehlbach BK, Chapotot F, Leproult R, Whitmore H, Poston J, Pohlman M, Miller A, Pohlman AS, Nedeltcheva A, Jacobsen JH, Hall JB, Van Cauter E. Temporal disorganization of circadian rhythmicity and sleep-wake regulation in mechanically ventilated patients receiving continuous intravenous sedation. Sleep. 2012 Aug 1;35(8):1105-14. doi: 10.5665/sleep.1998. PMID 22851806
- [Background] Huang HW, Zheng BL, Jiang L, Lin ZT, Zhang GB, Shen L, Xi XM. Effect of oral melatonin and wearing earplugs and eye masks on nocturnal sleep in healthy subjects in a simulated intensive care unit environment: which might be a more promising strategy for ICU sleep deprivation? Crit Care. 2015 Mar 19;19(1):124. doi: 10.1186/s13054-015-0842-8. PMID 25887528
- [Background] Hu RF, Jiang XY, Hegadoren KM, Zhang YH. Effects of earplugs and eye masks combined with relaxing music on sleep, melatonin and cortisol levels in ICU patients: a randomized controlled trial. Crit Care. 2015 Mar 27;19(1):115. doi: 10.1186/s13054-015-0855-3. PMID 25881268
- [Background] Kudchadkar SR, Aljohani OA, Punjabi NM. Sleep of critically ill children in the pediatric intensive care unit: a systematic review. Sleep Med Rev. 2014 Apr;18(2):103-10. doi: 10.1016/j.smrv.2013.02.002. Epub 2013 May 21. PMID 23702219
- [Background] Kudchadkar SR, Yaster M, Punjabi AN, Quan SF, Goodwin JL, Easley RB, Punjabi NM. Temporal Characteristics of the Sleep EEG Power Spectrum in Critically Ill Children. J Clin Sleep Med. 2015 Dec 15;11(12):1449-54. doi: 10.5664/jcsm.5286. PMID 26194730
- [Background] Oyarzun F. [Perception of a person's face and the process of personalization-depersonalization]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1985 Mar-Apr;13(2):74-6. No abstract available. Spanish. PMID 4061156
- [Background] Aitken LM, Rattray J, Hull A, Kenardy JA, Le Brocque R, Ullman AJ. The use of diaries in psychological recovery from intensive care. Crit Care. 2013 Dec 18;17(6):253. doi: 10.1186/cc13164. PMID 24351578
- [Background] Jones C, Backman C, Capuzzo M, Egerod I, Flaatten H, Granja C, Rylander C, Griffiths RD; RACHEL group. Intensive care diaries reduce new onset post traumatic stress disorder following critical illness: a randomised, controlled trial. Crit Care. 2010;14(5):R168. doi: 10.1186/cc9260. Epub 2010 Sep 15. PMID 20843344
- [Background] Kamdar BB, Yang J, King LM, Neufeld KJ, Bienvenu OJ, Rowden AM, Brower RG, Collop NA, Needham DM. Developing, implementing, and evaluating a multifaceted quality improvement intervention to promote sleep in an ICU. Am J Med Qual. 2014 Nov-Dec;29(6):546-54. doi: 10.1177/1062860613509684. Epub 2013 Nov 22. PMID 24270169
- [Background] Kamdar BB, Knauert MP, Jones SF, Parsons EC, Parthasarathy S, Pisani MA; Sleep in the ICU (SLEEPii) Task Force. Perceptions and Practices Regarding Sleep in the Intensive Care Unit. A Survey of 1,223 Critical Care Providers. Ann Am Thorac Soc. 2016 Aug;13(8):1370-7. doi: 10.1513/AnnalsATS.201601-087OC. PMID 27104770
- [Background] Benloucif S, Burgess HJ, Klerman EB, Lewy AJ, Middleton B, Murphy PJ, Parry BL, Revell VL. Measuring melatonin in humans. J Clin Sleep Med. 2008 Feb 15;4(1):66-9. PMID 18350967
- [Background] Curley MA, Harris SK, Fraser KA, Johnson RA, Arnold JH. State Behavioral Scale: a sedation assessment instrument for infants and young children supported on mechanical ventilation. Pediatr Crit Care Med. 2006 Mar;7(2):107-14. doi: 10.1097/01.PCC.0000200955.40962.38. PMID 16446601
- [Background] Franck LS, Harris SK, Soetenga DJ, Amling JK, Curley MA. The Withdrawal Assessment Tool-1 (WAT-1): an assessment instrument for monitoring opioid and benzodiazepine withdrawal symptoms in pediatric patients. Pediatr Crit Care Med. 2008 Nov;9(6):573-80. doi: 10.1097/PCC.0b013e31818c8328. PMID 18838937
- [Derived] Perry MA, Dawkins-Henry OS, Awojoodu RE, Blumenthal J, Asaro LA, Wypij D, Kudchadkar SR, Zuppa AF, Curley MAQ. Study protocol for a two-center test of a nurse-implemented chronotherapeutic restoring bundle in critically ill children: RESTORE Resilience (R2). Contemp Clin Trials Commun. 2021 Aug 19;23:100840. doi: 10.1016/j.conctc.2021.100840. eCollection 2021 Sep. PMID 34466711

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: RESTORE Resilience (R2), a 7-item individualized care bundle
Period: Overall Study
Arm/Group | Baseline | Intervention
Started | 20 | 36
Completed | 20 | 34
Not Completed | 0 | 2
Not completed — Withdrawn by parent/guardian | 0 | 1
Not completed — Withdrawn by physician | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline | Intervention | Total
Number analyzed (Participants) | 20 | 34 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 34 | 54
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.2 [1.0 to 12.0] | 5.3 [1.2 to 10.4] | 3.6 [1.1 to 10.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 14 | 20 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 18 | 33 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 13 | 22
  White | 8 | 17 | 25
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 34 | 54

OUTCOME MEASURES:

1. Primary Outcome: DARE (Daytime Activity Ratio Estimate), Post Extubation
Description: DARE = Daytime Activity Ratio Estimate after endotracheal extubation; DARE was calculated by dividing daytime (07:00-18:59) activity count by 24-hour activity count. A DARE of 50% indicates equal amount of activity between daytime and nighttime periods (loss of circadian rhythm), while a higher DARE indicates increased daytime activity and nighttime sleep consolidation.
Time Frame: From immediately after endotracheal extubation to PICU discharge, assessed for up to 28 days
Population: Primary outcome not available for 4 subjects.
Measure: Median (Inter-Quartile Range); unit: Percentage of total activity
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 18 | 32
Percentage of total activity | 56.7 [47.6 to 65.5] | 61.7 [52.7 to 64.8]

2. Secondary Outcome: Delta Between Average Nighttime and Average Daytime Salivary Melatonin Levels
Description: Delta between average nighttime (19:00 to 06:59) and average daytime (07:00 to 18:59) salivary melatonin levels
Time Frame: Day 5 of PICU hospitalization
Population: Data not available for all subjects.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 9 | 14
pg/mL | -16.4 [-28.0 to -0.1] | 0.1 [-5.9 to 7.5]

3. Secondary Outcome: Percentage of Study Days Where Light and Sound Were Modulated
Description: Percentage of study days where light and sound were modulated to reflect day-night variation in light and sound levels; 0 = no study days where light and sound were modulated; 100% = light and sound modulated on all study days
Time Frame: From date of enrollment until the date of PICU discharge, assessed for up to 28 days
Measure: Median (Inter-Quartile Range); unit: Percentage of study days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
Percentage of study days | 0 [0 to 0] | 100 [75 to 100]

4. Secondary Outcome: Percentage of Study Days Where the Patient Not Fed Enterally After Bedtime
Description: Percentage of study days where the patient was not fed enterally after bedtime
Time Frame: From date of enrollment until the date of PICU discharge, assessed for up to 28 days
Population: Data unavailable for all study subjects.
Measure: Median (Inter-Quartile Range); unit: Percentage of study days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 30
Percentage of study days | 43 [27 to 67] | 57 [38 to 100]

5. Secondary Outcome: Continuity in Nursing Care
Description: Continuity in Nursing Care Index (CINC) defined as (N nurses/N shifts)*100. Score range 0-100, lower scores are better.
Time Frame: From date of enrollment until the date of PICU discharge, assessed for up to 28 days
Measure: Median (Inter-Quartile Range); unit: units on a 0-100 scale
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
units on a 0-100 scale | 67 [52 to 77] | 67 [57 to 80]

6. Secondary Outcome: Pain Free Days
Description: Percentage of PICU days where pain was assessed (0-10 pain scale) without pain (Pain score <4)
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Population: Data not available for all subjects.
Measure: Median (Inter-Quartile Range); unit: Percentage of study days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 33
Percentage of study days | 80 [67 to 95] | 74 [45 to 86]

7. Secondary Outcome: Agitation Free Days
Description: Percentage of PICU days without agitation (Agitation = State Behavioral Scale [SBS; range -3 to +2] >/= 1)
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Measure: Median (Inter-Quartile Range); unit: Percentage of study days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
Percentage of study days | 55 [43 to 100] | 50 [25 to 75]

8. Secondary Outcome: Delirium Free Days
Description: Percentage of PICU days, where delirium was assessed, without delirium (using the CAPD, pCAM-ICU or psCAM-ICU; cut score determined by instrument)
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Population: Data not available for all subjects.
Measure: Median (Inter-Quartile Range); unit: Percentage of study days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 18 | 33
Percentage of study days | 74 [50 to 100] | 100 [60 to 100]

9. Secondary Outcome: Iatrogenic Withdrawal Syndrome (IWS) Free Days
Description: Percentage of PICU days without IWS (Withdrawal Assessment Tool - version 1 [WAT-1]; range of scores 0-12 where no IWS = WAT-1 < 3)
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Population: Subjects still in the PICU on day 5 or later.
Measure: Median (Inter-Quartile Range); unit: Percentage of study days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 15 | 26
Percentage of study days | 100 [100 to 100] | 100 [75 to 100]

10. Secondary Outcome: Peak Daily Dose of All Opioid Sedative Agents
Description: Highest daily mg/kg dose of all opioid sedative agents
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Measure: Median (Inter-Quartile Range); unit: mg/kg/day
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
mg/kg/day | 3.5 [1.7 to 6.1] | 2.9 [1.0 to 4.2]

11. Secondary Outcome: Cumulative Dose of All Opioid Sedative Agents
Description: Total PICU mg/kg dose of all opioid sedative agents received
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
mg/kg | 12.2 [4.6 to 23.5] | 7.6 [2.2 to 18.8]

12. Secondary Outcome: Total PICU Days of Opioid Sedation
Description: Total number of PICU days exposed to opioid sedation
Time Frame: From date of PICU admission until the date of PICU discharge, assessed for up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
days | 6 [5 to 11] | 7 [4 to 11]

13. Secondary Outcome: PICU Length of Stay
Description: Time between the start and stop of PICU care
Time Frame: From date and time of PICU admission until the date and time of PICU discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 34
days | 7.0 [4.1 to 15.3] | 7.1 [4.6 to 11.6]

14. Secondary Outcome: Parent Perception of Being well-cared-for
Description: Percent match on the 7-item family-centered care scale (FCCS); range from 0-100% match; where higher scores indicate a better match
Time Frame: On the date of PICU discharge, assessed once within an average of 2 weeks post PICU admission
Population: Data not available for all subjects.
Measure: Median (Inter-Quartile Range); unit: Percent Match
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 19 | 31
Percent Match | 100 [100 to 100] | 100 [86 to 100]

15. Secondary Outcome: DARE (Daytime Activity Ratio Estimate), Acute Phase
Description: as for outcome 1
Time Frame: From study enrollment to endotracheal extubation
Population: Data not available for all subjects.
Measure: Median (Inter-Quartile Range); unit: Percentage of total activity
Arm/Group | Baseline | Intervention
Number analyzed (Participants) | 20 | 33
Percentage of total activity | 53.3 [46.6 to 63.4] | 62.0 [55.3 to 65.1]

ADVERSE EVENTS:
Time Frame: From date of enrollment until the date of PICU discharge, assessed for up to 28 days
Arm/Group | Baseline | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/34
Other Adverse Events (participants affected / at risk) | 1/20 | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (N=20) | Intervention (N=34)
Extubation failure (reintubation within 24 hours) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Unplanned endotracheal tube extubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT04695392/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT04695392/ICF_001.pdf